CLINICAL TRIAL: NCT02562625
Title: Randomised Phase II Trial of Pembrolizumab and Radiotherapy in Melanoma
Brief Title: Trial of Pembrolizumab and Radiotherapy in Melanoma
Acronym: PERM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Recruitment
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4251
Record Dates: First submitted 2015-09-07; First posted 2015-09-29 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab Alone (Experimental): If the patient is randomised to the Pembrolizumab Arm Only then they will receive 200mg of pembrolizumab every 3 weeks.
  Interventions: Drug: Pembrolizumab
- Pembrolizumab plus Radiotherapy (Experimental): If The patient is randomised to this arm they will receive 200mg of pembrolizumab every 3 weeks in combination with a radiotherapy dosage of 24Gy in 3 fractions to be given over 3 consecutive days (only).
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Powder solution for infusion
Radiation: Radiotherapy — 24Gy
  Arms: Pembrolizumab plus Radiotherapy

SUMMARY:
Around 13,000 participants are diagnosed with melanoma in the UK each year and that number is growing quicker than any other cancer. About 20% of participants will see their cancer return following their initial treatment and at present would survive a median time of 912 months. In recent years, the development of new effective drugs has revolutionised the treatment of advanced melanoma, However, response rates are still low and new therapeutic approaches are needed.

This is a phase II study to look at the effectiveness and safety of the combination of a new drug called pembrolizumab plus radiotherapy compared to pembrolizumab alone. The purpose of this study is to see if the addition of radiotherapy to pembrolizumab is better than pembrolizumab alone by measuring how long these treatments can control the growth of the cancer. Also it will assess if by adding radiotherapy the investigators can see its effects not only in the tumour that has had radiotherapy but also in other tumours in the rest of the body.

DETAILED DESCRIPTION:
1. Risk and burden for participants Participants in this study have cancer but may still be eligible for standard therapy and may not show any benefit from the trial drug. If this is the case will be withdrawn from the trial and will receive standard care. The study itself carries a number of potential burdens:

   * Study drug and Radiotherapy. Although the dose and safety effects of the drug have been previously assessed in phase I trials and the radiotherapy used is considered standard of care, it is possible for participants to experience some side effects. To ensure any side effects are treated appropriately all participants will be reviewed regularly by experienced clinicians while having the study treatment. Comprehensive assessments for safety will be carried out.
   * Burden of frequent hospital visits and tests. Participants in this study must attend hospital every 3 weeks to check for any side effects of the drug, have routine blood and clinical biochemistry tests, clinical examinations and administer the next dose of pembrolizumab. Additionally, for research purposes some participants may consent to have additional tumour biopsies and blood tests. These will not be mandatory for all participants.
2. Recruitment Participants will be offered information about this study by their clinical teams if they are considered to meet the entry criteria and express interest in taking part in the study. It will be made clear that there will not necessarily be a therapeutic benefit from taking part in the study. It will also be made clear that, should participants decide not to take part their future care will not be affected. Participants will be given sufficient time and information to make an informed decision about entering the trial, all participants entering the trial will give written informed consent.
3. Confidentiality Participants will be linked to a unique identifier the code for which will be held on a password protected database held only by the study team. This study will run across twenty two hospital sites. Tumour data will be analysed at Manchester University and research blood will be analysed at Leeds University. Sample processing will take place using the trial ID only. No other patient identifiable information will be available on study samples. Investigators will have access to patient identifiable information on password protected NHS hospital notes and databases only.
4. Conflict of Interest Participants may be recruited to the study by those involved in their prior clinical care. Investigators do not expect conflict of interest between research and healthcare duties for a number of reasons: participants must give their full informed consent before entering the study, specifically regarding the unknown efficacy of the study drug. Those participants who do not continue in the study will maintain a relationship with the clinical team if required for symptom control. At the end of the study, participants will be able to access the results if they wish, through the Royal Marsden Website. They will also be sent a written summary of the results if they indicate this.
5. Use of tissue samples in future research If participants give their consent, any leftover blood or tissue samples which are not required for this study will be stored for future unspecified research in line with the human tissue act regulations. Access and use of samples for research purposes will require appropriate ethical approval. Future researchers will not be able to identify individual participants from their biobank data, demographic and clinical information will be available.

ELIGIBILITY:
INCLUSION

1. Be willing and able to provide written informed consent for the trial
2. Have a diagnosis of stage III (unresectable) or stage IV cutaneous melanoma or melanoma of unknown primary, as per AJCC staging system
3. Informed metastatic disease by diagnostic biopsy
4. Be more than 18 years of age on day of signing informed consent
5. Have at least one lesion and a maximum of 3 which are appropriate targets for high dose radiotherapy. This lesion must be 1cm-5cm in size and measurable by RECIST v1.1
6. Have in addition at least one other lesion which will not be irradiated but must be measurable by RECIST v1.1 to assess the abscopal effect of the treatment
7. Have a performance status of 0 or 1 on the ECOG performance scale

8. Demonstrate adequate organ function as defined in table 1 below. All screening labs should be performed within 7 days of randomisation

9 Female patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to randomisation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

10 Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year

11 Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

EXCLUSION

1. Has lesions that if irradiated would result in unacceptable radiation induced toxicity to normal tissue, in particular to the CNS and bowel
2. Requires palliative radiotherapy for symptom control
3. Is currently participating in or has participated in a study of an investigational agent or device within 4 weeks of the first dose of trial treatment
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
5. Has had a monoclonal antibody within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e. ≤Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
6. Has had chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤Grade 1 or at baseline) from adverse events due to a previously administered agent

   * Note: patients with an AE ≤Grade 2 neuropathy are an exception to this criterion and may qualify for the study
   * Note: if patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
7. Has history of severe colitis related to previous immunotherapy treatment
8. Has a known additional malignancy that is progressing or requires active treatment Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
10. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
11. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137
17. Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
18. Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected)
19. Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Objective: To evaluate if radiotherapy will enhance the efficacy of pembrolizumab in the treatment of patients with metastatic melanoma by induction of an abscopal effect. | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
  Evaluated by RECIST v1.1

OTHER OUTCOMES:
Evaluating response rates by RECIST v1.1 post treatment | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
  Evaluated by RECIST v1.1
Exploratory Objective: Identifying biomarkers that correlate with immunological response to therapy | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
  Assessed by immunohistochemistry analysis of tumour
Evaluating response in non-irradiated lesions | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
  Evaluated by RECIST criteria v1.1
Assessing the efficacy of pembrolizumab based on Progression Free Survival (PFS). | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
Assessing the efficacy of pembrolizumab based on Overall Survival (OS). | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
Assessing the safety and tolerability of pembrolizumab alone and in combination with high dose radiotherapy. | From date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 60 months
  Evaluated by RECIST criteria v1.1

CONTACTS AND LOCATIONS:
Overall Officials: James Dr Larkin, MD, Study Director — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden, London, United Kingdom